CLINICAL TRIAL: NCT02907073
Title: First In-human PET Imaging Studies With NIS Reporter [18F]BF4
Brief Title: Positron Emission Tomography (PET) Imaging Studies With NIS Reporter
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: pursuing IND
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Tim DeGrado, PI, Mayo Clinic
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-002494
Record Dates: First submitted 2016-09-13; First posted 2016-09-20 (Estimated); Results first posted 2019-05-17 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Myeloma; Endometrial Cancer
MeSH Terms: conditions — Neoplasms, Plasma Cell; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy Volunteers (Experimental): At the study visit, healthy subjects will have an initial physical exam, urine pregnancy test (if applicable) and will have catheters placed for i.v. drug administration and blood sampling. Vital signs, and blood samples will be obtained. Subjects will receive an infusion [18F]BF4 over 1 minute and PET imaging will begin. Three (3) PET/CT scanning procedures will be performed over a period of approximately 4 hours with two rest breaks in between. Venous blood samples for clinical laboratory tests will be taken before radiotracer administration and at 1.5 hours post-administration of radiotracer. In addition, venous blood samples will be taken during the PET/CT scans to determine blood pharmacokinetics and metabolite evaluation. Physical exam will be repeated at the end of the study.
  Interventions: Drug: BF4
- Myeloma patients (Experimental): For cancer patients undergoing virus treatments, subjects will undergo [18F]BF4-PET/CT imaging at baseline before virus administration and at day 9 following virus treatment. Subjects will be screened by physician specialists within their clinics. Subjects who qualify for the study will return to the clinic within 30 days of screening, have a urine pregnancy test (if applicable) and will have catheters placed for i.v. drug administration. Vital signs will be obtained. All subjects will then receive a single i.v. bolus of [18F]BF4 for injection and PET/CT imaging will begin. Biopsies will be performed to confirm NIS expression in tissue of tumor regions showing uptake of [18F]BF4 in up to three myeloma patients when the site is accessible for biopsy.
  Interventions: Drug: BF4
- Endometrial cancer patients (Experimental): For cancer patients undergoing virus treatments, subjects will undergo [18F]BF4-PET/CT imaging at baseline before virus administration and at day 9 following virus treatment. Subjects will be screened by physician specialists within their clinics. Subjects who qualify for the study will return to the clinic within 30 days of screening, have a urine pregnancy test (if applicable) and will have catheters placed for i.v. drug administration. Vital signs will be obtained. All subjects will then receive a single i.v. bolus of [18F]BF4 for injection and PET/CT imaging will begin. Biopsies will be performed to confirm NIS expression in tissue of tumor regions showing uptake of [18F]BF4 in up to three endometrial cancer patients when the site is accessible for biopsy.
  Interventions: Drug: BF4

INTERVENTIONS:
Drug: BF4 — Single IV dose of 9-11 millicurie (mCi) sodium [Fluorine-18] radiolabeled B4^F
  Other Names: Tetrafluoroborate, TFB

SUMMARY:
The goal of this proposal is to perform first-in-man evaluation of and experimental imaging agent F-18 tetrafluoroborate (BF4) or (TFB).

DETAILED DESCRIPTION:
F-18 tetrafluoroborate (BF4) or (TFB) is being used as a PET (Positron Emission Tomography) imaging biomarker for expression of the human sodium/iodide symporter (hNIS) in tissues. Imaging of functional hNIS activity in tissues with [18F]BF4 is anticipated to provide superior sensitivity and image quality to I-123 or Tc-99m SPECT for monitoring hNIS transduction effected by viral therapies. The proposed work is designed to 1) evaluate its safety, biodistribution, metabolism and radiation dosimetry characteristics in 8 healthy human volunteers and 2) evaluate the imaging feasibility in comparison with I-123 or Tc-99m SPECT of hNIS expression in a) 10 myeloma patients treated with Edmonston Measles virus-NIS (MV-NIS) and b) 10 endometrial cancer patients treated with vesicular stomatitis virus engineered to express human interferon and NIS (VSV-hINF-NIS). This data will be necessary to support future regulatory submissions.

ELIGIBILITY:
Inclusion Criteria:

* Four male and four female healthy volunteers, greater than 21 years of age.
* Subjects must provide written informed consent.
* Willingness to provide all biological specimens as required by the protocol

Exclusion Criteria:

Volunteers with any of the following are ineligible to enroll in this study:

* Have currently clinically significant cancer, neurologic, hepatic, renal, pulmonary, metabolic, or endocrine disturbances, especially thyroid disease;
* Current clinically significant cardiovascular disease. Clinically significant cardiovascular disease usually includes one or more of the following:

  1. cardiac surgery or myocardial infarction within the last 6 months;
  2. unstable angina;
  3. coronary artery disease that required a change in medication within the last 3 months;
  4. decompensated congestive heart failure;
  5. significant cardiac arrhythmia or conduction disturbance, particularly those resulting in atrial or ventricular fibrillation, or causing syncope, near syncope, or other alterations in mental status;
  6. severe mitral or aortic valvular disease;
  7. uncontrolled high blood pressure;
  8. congenital heart disease;
* History of drug or alcohol abuse within the last year, or prior prolonged history of abuse;
* Clinically significant infectious disease, including AIDS or HIV infection or previous positive test for hepatitis B, hepatitis C, HIV-1, or HIV-2;
* Women of childbearing potential must not be pregnant (negative urine Human Chorionic Gonadotropin (β-HCG) at the time of screen) or lactating over the course of the study. A commercial urine dipstick test will be performed within 48 hours prior to injection of [18F]BF4 unless the screening urine pregnancy test falls within 48 hours of injection.
* Volunteers who, in the opinion of the investigator, are otherwise unsuitable for a study of this type;
* History of severe drug allergy or hypersensitivity; or
* Volunteers who had received an investigational medication within the last 30 days or who have participated in a clinical trial with any experimental medication or radiopharmaceutical in the last 30 days. Additionally, the time between the last dose of the previous experimental medication and enrollment (completion of screening assessments) must be at least equal to 5 times the terminal half-life of the previous experimental medication.
* Volunteers who are taking drugs with narrow therapeutic windows, such as theophylline, or warfarin, heparin and other anticoagulant therapies

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-09; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy R DeGrado, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Volunteers: At the study visit, healthy subjects will have an initial physical exam, urine pregnancy test (if applicable) and will have catheters placed for i.v. drug administration and blood sampling. Vital signs, and blood samples will be obtained. Subjects will receive an infusion [18F]BF4 over 1 minute and Positron Emission Tomography (PET) imaging will begin. Three (3) PET/CT scanning procedures will be performed over a period of approximately 4 hours with two rest breaks in between. Venous blood samples for clinical laboratory tests will be taken before radiotracer administration and at 1.5 hours post-administration of radiotracer. In addition, venous blood samples will be taken during the PET/CT scans to determine blood pharmacokinetics and metabolite evaluation. Physical exam will be repeated at the end of the study.
  BF4: Single IV dose of 9-11 millicurie (mCi) sodium [Fluorine-18] radiolabeled B4^F
- Myeloma Patients: For cancer patients undergoing virus treatments, subjects will undergo [18F]BF4-PET/CT imaging at baseline before virus administration and at day 9 following virus treatment. Subjects will be screened by physician specialists within their clinics. Subjects who qualify for the study will return to the clinic within 30 days of screening, have a urine pregnancy test (if applicable) and will have catheters placed for i.v. drug administration. Vital signs will be obtained. All subjects will then receive a single i.v. bolus of [18F]BF4 for injection and PET/CT imaging will begin. Biopsies will be performed to confirm NIS expression in tissue of tumor regions showing uptake of [18F]BF4 in up to three myeloma patients when the site is accessible for biopsy.
  BF4: Single IV dose of 9-11 mCi sodium [Fluorine-18] radiolabeled B4^F
- Endometrial Cancer Patients: For cancer patients undergoing virus treatments, subjects will undergo [18F]BF4-PET/CT imaging at baseline before virus administration and at day 9 following virus treatment. Subjects will be screened by physician specialists within their clinics. Subjects who qualify for the study will return to the clinic within 30 days of screening, have a urine pregnancy test (if applicable) and will have catheters placed for i.v. drug administration. Vital signs will be obtained. All subjects will then receive a single i.v. bolus of [18F]BF4 for injection and PET/CT imaging will begin. Biopsies will be performed to confirm NIS expression in tissue of tumor regions showing uptake of [18F]BF4 in up to three endometrial cancer patients when the site is accessible for biopsy.
  BF4: Single IV dose of 9-11 mCi sodium [Fluorine-18] radiolabeled B4^F
Period: Overall Study
Arm/Group | Healthy Volunteers | Myeloma Patients | Endometrial Cancer Patients
Started | 8 | 0 | 0
Completed | 8 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated due to pursuing IND.
Groups:
- Healthy Volunteers: At the study visit, healthy subjects will have an initial physical exam, urine pregnancy test (if applicable) and will have catheters placed for i.v. drug administration and blood sampling. Vital signs, and blood samples will be obtained. Subjects will receive an infusion [18F]BF4 over 1 minute and PET imaging will begin. Three (3) PET/CT scanning procedures will be performed over a period of approximately 4 hours with two rest breaks in between. Venous blood samples for clinical laboratory tests will be taken before radiotracer administration and at 1.5 hours post-administration of radiotracer. In addition, venous blood samples will be taken during the PET/CT scans to determine blood pharmacokinetics and metabolite evaluation. Physical exam will be repeated at the end of the study.
  BF4: Single IV dose of 9-11 mCi sodium [Fluorine-18] radiolabeled B4^F
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteers | Myeloma Patients | Endometrial Cancer Patients | Total
Number analyzed (Participants) | 8 | 0 | 0 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (11) |  |  | 35 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 |  |  | 4
  Male | 4 |  |  | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0
  Asian | 3 |  |  | 3
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
  Black or African American | 0 |  |  | 0
  White | 5 |  |  | 5
  More than one race | 0 |  |  | 0
  Unknown or Not Reported | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 |  |  | 8

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Tissue Distribution of F-18 BF4 in Healthy Volunteers
Description: F-18 BF4 concentrations in major tissues (e.g., heart, blood pool, lung, liver, thyroid, stomach, kidney, brain, muscle) will be evaluated from the PET images from 0-240 minutes post-administration. Results will be used to compute radiation dosimetry estimates.
Time Frame: 0-240 minutes
Population: Outcome measures were performed in study arm of eight healthy volunteers. F or the myeloma and endometrial cancer arms of the study, the study was terminated due to pursuing Investigational New Drug application (IND).
Measure: Mean (Standard Deviation); unit: standardized uptake value (SUV)
Arm/Group | Healthy Volunteers | Myeloma Patients | Endometrial Cancer Patients
Number analyzed (Participants) | 8 | 0 | 0
standardized uptake value (SUV)
  Bone uptake - 2 h males | 0.8 (0.39) |  |
  Bone uptake - 2 h females | 1.4 (0.5) |  |
  Brain uptake - 2 h males | 0.39 (0.14) |  |
  Brain uptake - 2 h females | 0.42 (0.15) |  |
  Breast uptake - 2 h females | 2.8 (0.4) |  |
  Gallbladder uptake - 2 h males | 2.7 (1.5) |  |
  Gallbladder uptake - 2h females | 3.7 (1.0) |  |
  Intestinal uptake - 2h males | 2.9 (1.0) |  |
  Intestinal uptake - 2h females | 5.0 (2.7) |  |
  Kidney uptake - 2h males | 7.0 (2.5) |  |
  Kidney uptake - 2h females | 5.6 (0.7) |  |
  Liver uptake - 2h males | 2.3 (1.0) |  |
  Liver uptake - 2h females | 2.7 (0.5) |  |
  Lung uptake - 2h males | 1.0 (0.4) |  |
  Lung uptake - 2h females | 1.2 (0.4) |  |
  Muscle uptake - 2h males | 0.71 (0.31) |  |
  Muscle uptake - 2h females | 0.65 (0.35) |  |
  Myocardium - 2h males | 3.2 (0.9) |  |
  yocardium - 2h females | 2.8 (0.5) |  |
  Pancreas - 2h males | 3.4 (0.7) |  |
  Pancreas - 2h females | 3.1 (1.7) |  |
  Parotid gland - 2h males | 11 (9) |  |
  Parotid gland - 2h females | 20 (11) |  |
  Spleen - 2h males | 4.1 (1.2) |  |
  Spleen - 2h females | 4.3 (1.0) |  |
  Stomach - 2h males | 33 (15) |  |
  Stomach - 2h females | 72 (10) |  |
  Thyroid - 2h males | 55 (31) |  |
  Thyroid - 2h females | 50 (11) |  |

2. Secondary Outcome: Amount of Imaging Agent in Tumor (Uptake) in Myeloma and Endometrial Cancer Patients
Description: Areas of positive uptake within tumor, relative to background, measured by Standardized Update Value (SUV). PET SUV is tissue concentration/injected dose/body weight in grams.
Time Frame: Baseline, Day 9
Population: Healthy volunteers do not have tumors. The study in myeloma and endometrial cancer was terminated due to pursuing IND.
Arm/Group | Healthy Volunteers | Myeloma Patients | Endometrial Cancer Patients
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data collection was defined as 24 hours following last administration of study treatment.
Description: The study in eight healthy volunteers was completed. The study arms in myeloma and endometrial cancer were terminated due to pursuing IND.
Arm/Group | Healthy Volunteers | Myeloma Patients | Endometrial Cancer Patients
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/8 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated due to pursuing Investigational New Drug application (IND).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT02907073/Prot_SAP_000.pdf